CLINICAL TRIAL: NCT07188532
Title: Biologically-Adapted, Dose-Escalated Accelerated Radiotherapy for Ewing Sarcoma (BEAR)
Brief Title: Biologically-Adapted, Dose-Escalated Radiotherapy for the Treatment of Ewing Sarcoma, BEAR Trial
Acronym: BEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2411; NCI-2025-06507 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-004837 (Other: Mayo Clinic Institutional Review Board); BEAR (Other: Mayo Clinic Radiation Oncology); GMROR2411 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ewing Sarcoma; Round Cell Sarcoma With EWSR1-non-ETS Fusion
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Specimen Handling; Drug Therapy; Radiation; Congresses as Topic; Radiation Dose Hypofractionation; Magnetic Resonance Spectroscopy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Cohort A Group 1 (dose-escalated radiotherapy) (Experimental): Patients may receive SOC chemotherapy every 2 weeks for at least 3 cycles prior to radiotherapy. Patients then undergo hypofractionated or conventional dose-escalated radiotherapy daily, excluding weekends and holidays, for 25-36 treatment fractions in the absence of disease progression or unacceptable toxicity. Patients may also receive consolidation chemotherapy after completion of radiotherapy and/or surgical resection. Patients also undergo blood sample collection throughout the study. Additionally, patients may also undergo CT, PET/CT, and MRI with or without CT throughout the study at treating clinician's discretion.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Conventional Radiotherapy; Procedure: Definitive Surgical Resection; Radiation: Dose-escalated Radiation Therapy; Other: Electronic Health Record Review; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Cohort A Group 2 (standard dose radiotherapy) (Experimental): Patients may receive SOC chemotherapy every 2 weeks for at least 3 cycles prior to radiotherapy. Patients then undergo hypofractionated or conventional standard dose radiotherapy daily, excluding weekends and holidays, for 25-31 treatment fractions in the absence of disease progression or unacceptable toxicity. Patients may also receive consolidation chemotherapy after completion of radiotherapy and/or surgical resection. Patients also undergo blood sample collection throughout the study. Additionally, patients may also undergo CT, PET/CT, and MRI with or without CT throughout the study at treating clinician's discretion.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Conventional Radiotherapy; Procedure: Definitive Surgical Resection; Other: Electronic Health Record Review; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Cohort B (definitive radiotherapy, surgical resection) (Experimental): Patients may receive SOC chemotherapy every 2 weeks for at least 3 cycles prior to radiotherapy. Patients with tumor size < 8cm at diagnosis undergo definitive radiotherapy or surgical resection. Patients may also receive consolidation chemotherapy after completion of definitive radiotherapy or surgical resection. Patients also undergo blood sample collection throughout the study. Additionally, patients may also undergo CT, PET/CT, and MRI with or without CT throughout the study at treating clinician's discretion.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Definitive Surgical Resection; Other: Electronic Health Record Review; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Cohort C (radiotherapy, surgical resection) (Experimental): Patients may receive SOC chemotherapy every 2 weeks for at least 3 cycles prior to radiotherapy. Patients undergo radiotherapy before or after undergoing definitive surgical resection. Patients may also receive consolidation chemotherapy after completion of definitive radiotherapy and surgical resection. Patients also undergo blood sample collection throughout the study. Additionally, patients may also undergo CT, PET/CT, and MRI with or without CT throughout the study at treating clinician's discretion.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Conventional Radiotherapy; Procedure: Definitive Surgical Resection; Other: Electronic Health Record Review; Radiation: External Beam Radiation Therapy; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Chemotherapy — Given chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Conventional Radiotherapy — Undergo conventional radiotherapy
  Other Names: 2-Dimensional Conventional Radiation Therapy; 2D Conventional Radiotherapy; 2D Radiotherapy; 2D-RT; Radiation, 2D Conventional
  Arms: Cohort A Group 1 (dose-escalated radiotherapy); Cohort A Group 2 (standard dose radiotherapy); Cohort C (radiotherapy, surgical resection)
Procedure: Definitive Surgical Resection — Undergo definitive surgical resection
Radiation: Dose-escalated Radiation Therapy — Undergo hypofractionated or conventional radiotherapy
  Other Names: Dose-escalated RT
  Arms: Cohort A Group 1 (dose-escalated radiotherapy)
Other: Electronic Health Record Review — Ancillary studies
Radiation: External Beam Radiation Therapy — Undergo definitive radiotherapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
  Arms: Cohort B (definitive radiotherapy, surgical resection); Cohort C (radiotherapy, surgical resection)
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
  Arms: Cohort A Group 1 (dose-escalated radiotherapy); Cohort A Group 2 (standard dose radiotherapy); Cohort C (radiotherapy, surgical resection)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo hypofractionated or conventional standard radiotherapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Cohort A Group 2 (standard dose radiotherapy); Cohort C (radiotherapy, surgical resection)

SUMMARY:
This clinical trial evaluates the effect of radiotherapy doses based on tumor size and tumor-specific characteristics (biologically-adapted) in treating patients with Ewing sarcoma. Radiotherapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Conventional radiotherapy uses minimal imaging support to determine the positioning of radiotherapy. Hypofractionated radiotherapy delivers higher doses of radiotherapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Dose-escalated radiotherapy uses doses that are higher than those used in conventional radiotherapy. Larger tumor sizes and other tumor-specific characteristics have been shown to be related to poorer outcomes. In addition, after dose-escalated radiotherapy, patients with larger tumors have demonstrated improved control of the disease at the primary tumor site. Giving biologically-adapted, dose-escalated radiotherapy may reduce the return of the cancer at the primary tumor site in patients with Ewing sarcoma with large tumors and other unfavorable characteristics. This clinical trial also evaluates the role of biomarkers in patients with Ewing sarcoma. Studying samples of blood and tumor tissue from patients with Ewing sarcoma in the laboratory may help doctors learn more about predicting the amount of disease and the likelihood of the cancer coming back.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION: INCLUSION CRITERIA

* Histological confirmation of Ewing sarcoma, including both skeletal and extra-skeletal primary tumors. Patients with "Ewing-like" sarcoma may be eligible if patients are planned to be treated per Ewing treatment paradigms, as defined in this clinical trial REGISTRATION: INCLUSION CRITERIA
* Patients of age ≥ 2 years are eligible for the study
* Lansky or Karnofsky performance status ≥ 70
* Ability to provide written informed consent and complete questionnaire(s) by themselves or with assistance
* Willing to provide blood samples for correlative research purposes
* COHORT A ONLY: Willing to provide biopsy sample to run Mayo Complete Solid Tumor Panel

Exclusion Criteria:

REGISTRATION: EXCLUSION CRITERIA

* Prior chemotherapy or radiotherapy that, in the opinion of the treating medical oncologist or radiation oncologist, is considered to interfere with the current treatment or measurement of outcomes
* Receiving any investigational agent which would be considered as a treatment for the primary neoplasm that is considered by the investigator to interfere with the current treatment or measurement of outcomes

  * Note: Co-enrollment on another clinical trial is allowed per the treating radiation oncologist's discretion
* Other active malignancy ≤ 1 year prior to registration that is considered by the investigator to interfere with the current treatment or measurement of outcomes
* Patients that have severe co-morbid systemic illness or other disease which would interfere significantly with the current treatment or measurement of outcomes
* Patients that have active uncontrolled systemic infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric illness or social situation that would limit study adherence
* Any of the following:

  * Pregnant patients
  * Nursing patients

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in local failure for patients with large tumors (Cohort A) | Up to 2 years
  Large tumors defined as ≥ 8cm. Will be compared to the historical control of 14.3%. Local failure will be defined per the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Incidence of targeted, late grade 3 or greater adverse events (Cohort A) | Up to 1 year after completion of local therapy
  Assessed per RECIST version 1.1.
Event-free survival (Cohort A) | Up to 1 year after completion of local therapy
  Event-free survival (EFS) is defined as the time from study entry to any progression of disease or recurrence of disease or death from any cause, whichever occurs first.
Time to progression (Cohort A) | Up to 1 year after completion of local therapy
  Will be calculated descriptively, via frequencies and percentages at various timepoints of interest, including the 1-year local control rate.
Overall survival (Cohort A) | Up to 1 year after completion of local therapy
  Overall survival (OS) is defined as the time from study entry to death from any cause, estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Roman O. Kowalchuk, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials